CLINICAL TRIAL: NCT01128270
Title: Pharmacotoxicology of Trichloroethylene Metabolites Aim 3
Brief Title: Pharmacotoxicology of Trichloroethylene Metabolites
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#107-10; RO1ESO141617 (Other Grant/Funding Number: National Institute of Health RO1ESO14167)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Dichloroacetate; Chloral Hydrate; Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1A: Chloral Hydrate and DCA: Env (Experimental): Subjects consume Chloral Hydrate 1.5ug/kg by mouth for 5 nights. On the 6th day they consume DCA 2.5ug/kg by mouth and have blood samples drawn. (Period 1)
  Interventions: Drug: Dichloroacetate environmental dose; Drug: Chloral Hydrate environmental dose
- 1B: Chloral Hydrate Env dose (Experimental): Drug Study Subjects are admitted to the clinical research unit and receive 1.5 ug/kg (environmental dose) of Chloral Hydrate for 5 nights. Pharmacokinetics are done on days 1 and day 5. (Period 2)
  Interventions: Drug: Chloral Hydrate environmental dose
- 2A: Chloral Hydrate and DCA therapeutic (Experimental): Drug Study Subjects are admitted to the clinical research center and receive a clinical dose of Chloral Hydrate for 5 nights (25mg/kg). On day 6 they are given a clinical dose (25mg/kg)of Dichloroacetate. (Period 3)
  Interventions: Drug: Dichloroacetate therapeutic dose; Drug: Chloral Hydrate therapeutic dose
- 2B: Chloral Hydrate Therapeutic (Experimental): Subjects are given 25 mg/kg of Chloral Hydrate for five nights. Pharmacokinetics are done on days 1 and 5. (Period 4)
  Interventions: Drug: Chloral Hydrate therapeutic dose

INTERVENTIONS:
Drug: Dichloroacetate environmental dose — On day 6 they receive Dichloroacetate 2.5 ug/kg orally times 1 and have pharmacokinetics.
  Other Names: DCA
  Arms: 1A: Chloral Hydrate and DCA: Env
Drug: Chloral Hydrate environmental dose — Study subjects are given 1.5 ug/kg of Chloral Hydrate for 5 nights and pharmacokinetics are done on night 1 and 5.
  Arms: 1A: Chloral Hydrate and DCA: Env; 1B: Chloral Hydrate Env dose
Drug: Dichloroacetate therapeutic dose — Subjects receive 25 mg/kg DCA on Day 6. Pharmacokinetics are done on nights 1 and nights 5.
  Other Names: DCA
  Arms: 2A: Chloral Hydrate and DCA therapeutic
Drug: Chloral Hydrate therapeutic dose — Subject is given 25 mg/kg of Chloral Hydrate for five nights.
  Arms: 2A: Chloral Hydrate and DCA therapeutic; 2B: Chloral Hydrate Therapeutic

SUMMARY:
This is a research study to look at how Dichloroacetate (DCA), and investigational drug and chloral hydrate are broken down in the body. The purpose of the study is to better understand how humans metabolize these two common chemicals that are widely present in the environment. The study focuses on how the drug chloral hydrate is broken down and how it effects DCA

DETAILED DESCRIPTION:
The subject's general health is assessed by a history and physical exam and routine blood work. I normal the individual undergoes five nights of receiving 1.5ug/kg of chloral hydrate. On day 6 the individual receives 2.5 micrograms/kg of Dichloroacetate (DCA) and kinetics are drawn. After 30 days the subject comes back and receives 1.5ug/kg of chloral hydrate for five nights and has kinetics drawn on night one and five. On days 6-9 the subject returns for a blood draw. After 30 days the same process as above is done except the subject receives 1gram of chloral hydrate for five nights and 25mg/kg of Dichloroacetate one day then 30 days later the subject receives 1gram of chloral hydrate for five nights and has kinetics done on night one and five and blood samples drawn on days 6-9

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal screening labs

Exclusion Criteria:

* no gastrointestinal surgery
* no smoking
* no medication
* not pregnant

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Medicine, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited using an ad approved by the Institutional Review Board (IRB) and by undergoing a screening exam to determine eligibility.
Pre-assignment Details: There were 27 total participants, with 4 eligible sessions (periods) for each, with the order to be randomized. As per CT.Gov instructions, the periods are identified by treatment rather than order.There were no planned comparisons between the arms of this pharmacological study. Withdrawals entered but did not reach baseline.
Groups:
- All Subjects: The intent was to have all subjects participate in all four sessions (periods). These were environmental chloral hydrate +/- environmental DCA and therapeutic chloral hydrate +/- therapeutic DCA. Patient participation: 4 Sessions (N=2), 3 Sessions (N=1), 2 Sessions (N=6), 1 Session (N=8), 0 Sessions (N=10), Total: N=27 patients participated in 31 sessions.
Period: Environment Chloral Hydrate and DCA (1A)
Arm/Group | All Subjects
Started | 7
Completed | 7
Not Completed | 0
Period: Environmental Chloral Hydrate (1B)
Arm/Group | All Subjects
Started | 8 (Per the suggestion from Heather, periods are not in chronological order, but defined by treatment.)
Completed | 8
Not Completed | 0
Period: Therapeutic Chloral Hydrate and DCA (2A)
Arm/Group | All Subjects
Started | 8
Completed | 8
Not Completed | 0
Period: Therapeutic Chloral Hydrate (2B)
Arm/Group | All Subjects
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Withdrawals before their treatment was to begin, as all were scheduled to participate in all 4 participate.
Groups:
- All Subjects: Intent was to have all subjects participate in all sessions (periods)
Arm/Group | All Subjects
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Plasma DCA (Microgram/ml) After 5 Days of Therapeutic Level Chloral Hydrate on Arm 2A.
Description: After 5 days of of therapeutic level Chloral Hydrate, the levels of Dichloroacetate in the plasma were measured.
Time Frame: 6 Days
Measure: Mean (Standard Deviation); unit: micrograms/ml
Groups:
- Therapeutic Chloral Hydrate and DCA (2A): Arm 2A: Subjects are given Chloral Hydrate (25 mg/kg for five nights) and therapeutic Dichloroacetate on Day 1 (25 mg/Kg.) Pharmacokinetics are done on days 1 and 5. This outcome only applies to Period 3.
Arm/Group | Therapeutic Chloral Hydrate and DCA (2A)
Number analyzed (Participants) | 8
micrograms/ml | 1.64 (0.40)
Statistical Analysis 1: Comparison: Therapeutic Chloral Hydrate and DCA (2A); No comparison is relevant. The statistical method is how we obtained the point estimate and confidence interval. No test was intended; Test type: Superiority or Other; Analysis applies only to Arm 2A. (Period 3); Mean of one group (2A) = 1.64, 95% CI 2-sided [1.31 to 1.97], Standard Deviation 0.40 — Only arm 2A is relevant to this variable. There is no intended statistical comparison, but the point estimate for the mean level and 95% confidence interval are provided

2. Primary Outcome: Difference in Half Lives 5 Day Less One Day Exposure in Trichloroacetate
Description: Elimination Half-life Difference on Arm 2B for 13C-Labeled trichloroacetate between day 5 (prolonged exposure) and day 1 (de novo exposure) after therapeutic level exposure to Chloral Hydrate. This outcome only applies to Period 4. Trichloroacetate is a marker, not an intervention.
Time Frame: 5 days
Population: This applies only to Arm 2B (Therapeutic Chloral Hydrate without DCA.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Therapeutic Chloral Hydrate (2B): Arm 2B: Subjects are given Chloral Hydrate (25 mg/kg for five nights)(25 mg/Kg.) Pharmacokinetics are done on days 1 and 5.
Arm/Group | Therapeutic Chloral Hydrate (2B)
Number analyzed (Participants) | 8
minutes | 2432 (1403)
Statistical Analysis 1: Comparison: Therapeutic Chloral Hydrate (2B); Only relevant to Arm 2B; Test type: Superiority or Other; p = 0.0017, t-test, 2 sided; Mean Difference (Net) = 2432, 95% CI 2-sided [1260 to 3606], Standard Deviation 1403

3. Primary Outcome: Urinary Maleylacetone Levels After 5 Day Exposure to Therapeutic Chloral Hydrate (Arm 2B)
Description: The levels were clinically indetectable at baseline and the question was whether or not substantive levels would be noted at after 5 days exposure to Chloral Hydrate. Detectable, but low levels were detected.
Time Frame: 5 days
Population: all eligible participants to arm 2B (Period 4)
Measure: Mean (Standard Deviation); unit: micrograms per ml clorohydrate
Arm/Group | Therapeutic Chloral Hydrate (2B)
Number analyzed (Participants) | 8
micrograms per ml clorohydrate | 0.38 (0.17)
Statistical Analysis 1: Comparison: Therapeutic Chloral Hydrate (2B); Only relevant for arm 2B; Test type: Superiority or Other; Mean = 0.38, 95% CI 2-sided [0.24 to 0.51], Standard Deviation 0.17

4. Secondary Outcome: Detectable DCA After Day 1 in Serum (0=No 1=Yes)
Description: All four arms receive Chloral Hydrate on Day 1 (arms 1A and 1B environmental levels) and (arms 2A and 2B therapeutic levels). The question is could Dichloroacetate be detected in serum at the end of day 1. This analysis is purely descriptive, and no comparisons were planned.
Time Frame: 1 day
Population: All eligible session completers
Measure: Number; unit: participants
Groups:
- Environmental Chloral Hydrate and DCA (1A): Arm 1A: Subjects are given Chloral Hydrate (1.5mcg/kg for five nights) and environmental Dichloroacetate on Day 1 (2.5 mcg/Kg.)pharmacokinetics are done on days 1 and 5.
- Environmental Chloral Hydrate (1B): Arm 1B: Subjects are given Chloral Hydrate (1.5mcg/kg for five nights). Pharmacokinetics are done on days 1 and 5.
- Therapeutic Chloral Hydrate and DCA (2A): Arm 2A: Subjects are given Chloral Hydrate (25 mg/kg for five nights) and therapeutic Dichloroacetate on Day 1 (25 mg/Kg.) Pharmacokinetics are done on days 1 and 5.
Arm/Group | Environmental Chloral Hydrate and DCA (1A) | Environmental Chloral Hydrate (1B) | Therapeutic Chloral Hydrate and DCA (2A) | Therapeutic Chloral Hydrate (2B)
Number analyzed (Participants) | 7 | 8 | 8 | 8
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for an average of 2 years.
Groups:
- 1A: Chloral Hydrate+DCA (Environmental): This is Period 1. See description of periods for full details.
- Chloral Hydrate (Environmental): This is Period 2. See description of periods for full details.
- Chloral Hydrate +DCA (Therapeutic Dose): This is Period 3. See description of periods for full details.
- Chloral Hydrate (Therapeutic Dose): This is Period 4 See description of periods for full details.
Arm/Group | 1A: Chloral Hydrate+DCA (Environmental) | Chloral Hydrate (Environmental) | Chloral Hydrate +DCA (Therapeutic Dose) | Chloral Hydrate (Therapeutic Dose)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/7 | 3/8 | 2/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Chloral Hydrate+DCA (Environmental) (N=7) | Chloral Hydrate (Environmental) (N=8) | Chloral Hydrate +DCA (Therapeutic Dose) (N=8) | Chloral Hydrate (Therapeutic Dose) (N=8)
Abdominal cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated liver enzymes (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
High Blood Pressure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Subjects were asked to wait 30 days in between doses of medication. Some of the participants could not wait the entire 4 months to finish the study and thus dropped out before they completed the 4 arms. Ten were enrolled, screened, but did not start

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No